CLINICAL TRIAL: NCT01119638
Title: Post Marketing Study of Escitalopram Versus Risperidone for the Treatment of Behavioral and Psychological Symptoms Amongst Alzheimer's Disease Patients
Brief Title: Escitalopram Treatment for BPSD in Alzheimer's Disease in Comparison to Risperidone
Acronym: EscBPSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abarbanel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Yoram Barak, Director of Psychogeriatrics, Abarbanel Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABR-BPSD-001; CO01ABR01022008 (Other Grant/Funding Number: Lundbeck A/S)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Agitation; Psychosis; Alzheimer's Disease
Keywords: Alzheimer's disease; BPSD; escitalopram; Risperidone; Agitation; Psychosis; Dementia; Elderly
MeSH Terms: conditions — Psychomotor Agitation; Psychotic Disorders; Alzheimer Disease; Dementia | interventions — Escitalopram; Dexetimide; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram Drug (Active Comparator): Drug:
  Patients in the escitalopram group will receive 5 mgs/d for the first week and than 10 mgs/d till completion.
  Interventions: Drug: Escitalopram
- Risperidone Drug (Active Comparator): Patients in the risperidone group will receive 0.5 mgs/d for the first week and than 1.0 mg/d till completion.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Escitalopram — Patients in the escitalopram group will receive 5 mgs/d for the first week and than 10 mgs/d till completion.
  Other Names: Cipralex
  Arms: Escitalopram Drug
Drug: Risperidone — Patients in the risperidone group will receive 0.5 mgs/d for the first week and than 1.0 mg/d till completion.
  Other Names: Risperdal
  Arms: Risperidone Drug

SUMMARY:
Behavioral and psychological symptoms of dementia (BPSD) are among the most distressing manifestations of dementia. Pharmacotherapy is frequently used and especially in institutional settings. Current guidelines recommend the use of second-generation antipsychotics (SGAs). Nonetheless, there are concerns regarding both their safety and effectiveness in patients with dementia. Inconclusive evidence support the use of other psychoactive agents such as SSRI antidepressants or cognitive enhancers.

In two published studies citalopram was as efficacious as, but better tolerated than perphenazine or risperidone in patients with BPSD.

Thus, with proven efficacy and a beneficial safety profile the evaluation of the use of escitalopram for BPSD is warranted.

DETAILED DESCRIPTION:
Behavioral and psychological symptoms of dementia (BPSD) as agitation or psychosis are among the most distressing manifestations of dementia. The evidence-based management of these symptoms includes the search for treatable physical and environmental precipitants, support and psychoeducation for primary caregivers and psychosocial interventions. Nevertheless, pharmacotherapy is frequently used and especially in institutional settings. Current guidelines recommend the use of second-generation antipsychotics (SGAs). Nonetheless, there are concerns regarding both their safety and effectiveness in patients with dementia. Recent research has resulted in a 'black-box" warning concerning the safety of using SGAs for BPSD. Sparse and inconclusive evidence support the use of other psychoactive agents such as SSRI antidepressants or cognitive enhancers.

In two published randomized controlled trials, citalopram was more efficacious than placebo and as efficacious as, but better tolerated than perphenazine or risperidone in patients with dementia hospitalized for the treatment of agitation or psychosis.

Thus, with proven efficacy and a beneficial safety profile the evaluation of the use of escitalopram for BPSD is warranted.

A 6-week parallel groups, randomized, controlled trial in patients with dementia hospitalized because of behavioral symptoms will be conducted at the Abarbanel MHC.

Participants will be consecutively recruited on an inpatient unit. Randomization will be based on a table of random numbers held centrally by an uninvolved physician.

The study will be of a "double-blind" design. All medications in identical packaging will be distributed to the ward from a central pharmacy.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will fulfill criteria for dementia of the Alzheimer's type (according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition). The score on the Mini-Mental State Examination (MMSE) has to be between 5 and 26.

Eligible patients will suffer from delusions, hallucinations, aggression, or agitation that developed after the onset of dementia and is severe enough to disrupt their functioning and, in the opinion of the study physicians, to justify treatment with antipsychotic drugs.

Signs and symptoms of psychosis, aggression, or agitation will have to occur nearly daily during the week prior to enrollment.

A frequency rating of "often" or "more frequently" and a severity rating of at least "moderate" are required for delusions, hallucinations, agitation, or "aberrant motor behavior" in the Neuropsychiatric Inventory (NPI).

Exclusion Criteria:

Patients will be excluded if they had received a diagnosis of a primary psychotic disorder (e.g., schizophrenia), delirium, other dementia. Patients will also be excluded if they were going to receive treatment with a cholinesterase inhibitor or antidepressant medication, had previously been treated with escitalopram for BPSD, or had contraindications to the two study drugs.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in total score on the NPI. | from first treatment to end of study at 6 weeks

SECONDARY OUTCOMES:
Time from initial treatment to the discontinuation of treatment for any reason. | time to discontinuation for any reason
  we shall consider any reason for stopping the study medications to be avalid reason for "discontinuation. This measure was deemed important by the NIH for dementia drug studies.

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Barak, MD, MHA, Principal Investigator — Abarbanel MHC, Israel.
Locations (1):
- Abarbanel MHC, Bat Yam, Israel

REFERENCES:
- [Background] Pollock BG, Mulsant BH, Rosen J, Mazumdar S, Blakesley RE, Houck PR, Huber KA. A double-blind comparison of citalopram and risperidone for the treatment of behavioral and psychotic symptoms associated with dementia. Am J Geriatr Psychiatry. 2007 Nov;15(11):942-52. doi: 10.1097/JGP.0b013e3180cc1ff5. Epub 2007 Sep 10. PMID 17846102